CLINICAL TRIAL: NCT03890536
Title: Intestinal Microbiome Composition in Infants With Biliary Atresia
Brief Title: Intestinal Microbiome Composition in Infants With Biliary Atresia (BA)
Acronym: BA
Status: Withdrawn | Type: Observational
Why Stopped: Study never began enrolling. Study team left institution.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: CIN001-Microbiome study in BA
Record Dates: First submitted 2019-01-30; First posted 2019-03-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Biliary Atresia; Intrahepatic Cholestases; Normal Controls
Keywords: Microbiome
MeSH Terms: conditions — Biliary Atresia; Cholestasis, Intrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool specimens will be collected from infants with Biliary atresia, non-biliary atresia liver disease and control subjects with no disease. Bacterial genomic DNA will be isolated from stool samples of the above-mentioned subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biliary atresia: Biliary atresia is an obstructive cholangiopathy of infancy. It is the most common cause of neonatal cholestasis and the most frequent indication for liver transplantation in children. Patients with biliary atresia have conjugated hyperbilirubinemia (serum direct bilirubin > 1mg/dL) AND are scheduled for/undergo exploratory laparotomy for diagnosis and Kasai portoenterostomy for surgical treatment of BA.
- Non-BA=disease controls: All infants with other cholestatic syndromes (except biliary atresia) will be eligible for study enrollment in disease controls/non-biliary atresia. This involves the diagnosis of liver diseases caused by syndromes of intrahepatic cholestasis with or without hyperbilirubinemia.
- Normal: All healthy infants with no acute or chronic liver related illness.

SUMMARY:
A prospective observational study in infants with biliary atresia and controls to determine whether the composition of the intestinal microbiome is specific for biliary atresia will be conducted.

The hypothesis of the study is "infants with biliary atresia have a unique microbiome signature at the time of diagnosis and changes in population dynamics occur during disease progression". The microbiome will be determined at diagnosis and at well-defined time points during the natural history of the disease.

DETAILED DESCRIPTION:
Biliary atresia, the most common cause of neonatal cholestasis, results from a fibrosing and inflammatory obstruction of extrahepatic bile ducts of unknown etiology. Infants with neonatal cholestasis will be enrolled at the time of diagnosis. Those that undergo exploratory laparotomy and are diagnosed with biliary atresia will form the "biliary atresia".

The development of the normal bacterial flora is a dynamic process that varies in early postnatal ages and may be influenced by disease states. To control for age differences, the composition of the microbiome in subjects with other causes of neonatal liver diseases (non-biliary atresia or disease-controls) and age-matched healthy subjects (normal controls) will be determined.

Subjects with biliary atresia will be enrolled at diagnosis, at which time a stool sample and a 2 mL blood sample will be obtained. Thereafter, a stool sample will be obtained at 3±1 months after hepatoportoenterostomy (HPE) and at 24±6 months of age. A stool sample and a 2 ml blood sample will also be obtained if/when subjects are admitted to the hospital for an evaluation and treatment of presumed infection (example: ascending cholangitis) and at the time of liver transplantation.

Similar samples will also be obtained from healthy subjects (normal controls) and patients diagnosed with other cholestatic syndromes (non-biliary atresia or disease-controls) at ages that match those of subjects with biliary atresia. Samples will be used for bacterial DNA isolation, which will be used for bacterial and mammalian gene sequencing using next-generation sequencing methods, followed by statistical analysis to identify unique microbiome compositions or alterations that are associated with particular disease (biliary atresia or non-BA controls) or clinical outcomes including response to HPE, ascending cholangitis and progression of liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   -Birth to 5 months
2. Disease state: Must meet either (a), (b), or (c) for eligibility.

   a) Biliary atresia:
   * Conjugated hyperbilirubinemia (serum direct bilirubin > 1mg/dL) AND demonstration of obstruction of extra hepatic bile ducts by examination of histological sections of extra hepatic bile ducts

     b) Neonatal cholestasis secondary to other causes of liver disease:
   * Diagnosis of liver disease caused by syndromes of intrahepatic cholestasis with or without hyperbilirubinemia

     c) Normal controls:
   * No acute or chronic liver related illness
3. Signed informed consent/assent

Exclusion Criteria:

1. Evidence of multi-organ system failure (e.g. combined liver and kidney failure)
2. For subjects < 5 months old, treatment with antibiotics prior to enrollment into study

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Biliary atresia, the most common cause of neonatal cholestasis, results from a fibrosing and inflammatory obstruction of extrahepatic bile ducts of unknown etiology. Infants with neonatal cholestases due to other causes and age-matched healthy controls will be enrolled.
  This is a prospective study that starts at the time of evaluation of neonatal cholestasis and will collect samples and clinical data during the progression of liver disease. A subject will be eligible for study once it is determined that the subject meets entry criteria either into the study or disease-control cohorts or the normal control cohort.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Change in intestinal microbiome signature. | Through study completion, an average of 24 months.
  Change in intestinal microbiome signature at the time of diagnosis of biliary atresia (up to 3 months of age/ at HPE) as compared with disease control and normal.

SECONDARY OUTCOMES:
Microbiome signature and serum direct/ conjugated bilirubin. | Through study completion, an average of 24 months.
  Correlation between the microbiome signature and normalization of serum direct/ conjugated bilirubin 3months after HPE.
Microbiome signature and survival at 1 yr of age. | Through study completion, an average of 36 months.
  Correlation between the microbiome signature and survival with the native liver at 1 yr of age.
Microbiome signature and survival at 2 yr of age. | Through study completion, an average of 48 months.
  Correlation between the microbiome signature and survival with the native liver at 2 yr of age.
Microbiome signature and ascending cholangitis. | Through study completion, an average of 48 months.
  Change in intestinal microbiome signature specific for ascending cholangitis up to and include 2 yr of age.
Change in microbiome signature and liver transplant. | Through study completion, an average of 48 months.
  Change in microbiome signature specific for end-stage liver disease (liver transplant) up to and include 2 yr of age..

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Bezerra, MD, Principal Investigator — Professor of Pediatrics
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balistreri WF, Grand R, Hoofnagle JH, Suchy FJ, Ryckman FC, Perlmutter DH, Sokol RJ. Biliary atresia: current concepts and research directions. Summary of a symposium. Hepatology. 1996 Jun;23(6):1682-92. doi: 10.1002/hep.510230652. PMID 8675193
- [Background] Bessho K, Bezerra JA. Biliary atresia: will blocking inflammation tame the disease? Annu Rev Med. 2011;62:171-85. doi: 10.1146/annurev-med-042909-093734. PMID 21226614
- [Background] Mack CL, Feldman AG, Sokol RJ. Clues to the etiology of bile duct injury in biliary atresia. Semin Liver Dis. 2012 Nov;32(4):307-16. doi: 10.1055/s-0032-1329899. Epub 2013 Feb 8. PMID 23397531
- [Background] Mouzaki M, Comelli EM, Arendt BM, Bonengel J, Fung SK, Fischer SE, McGilvray ID, Allard JP. Intestinal microbiota in patients with nonalcoholic fatty liver disease. Hepatology. 2013 Jul;58(1):120-7. doi: 10.1002/hep.26319. Epub 2013 May 14. PMID 23401313
- [Background] Tabibian JH, Talwalkar JA, Lindor KD. Role of the microbiota and antibiotics in primary sclerosing cholangitis. Biomed Res Int. 2013;2013:389537. doi: 10.1155/2013/389537. Epub 2013 Oct 22. PMID 24232746
- [Background] Kane M, Case LK, Kopaskie K, Kozlova A, MacDearmid C, Chervonsky AV, Golovkina TV. Successful transmission of a retrovirus depends on the commensal microbiota. Science. 2011 Oct 14;334(6053):245-9. doi: 10.1126/science.1210718. PMID 21998394
- [Background] Kuss SK, Best GT, Etheredge CA, Pruijssers AJ, Frierson JM, Hooper LV, Dermody TS, Pfeiffer JK. Intestinal microbiota promote enteric virus replication and systemic pathogenesis. Science. 2011 Oct 14;334(6053):249-52. doi: 10.1126/science.1211057. PMID 21998395
- [Background] Schloss PD, Westcott SL, Ryabin T, Hall JR, Hartmann M, Hollister EB, Lesniewski RA, Oakley BB, Parks DH, Robinson CJ, Sahl JW, Stres B, Thallinger GG, Van Horn DJ, Weber CF. Introducing mothur: open-source, platform-independent, community-supported software for describing and comparing microbial communities. Appl Environ Microbiol. 2009 Dec;75(23):7537-41. doi: 10.1128/AEM.01541-09. Epub 2009 Oct 2. PMID 19801464